CLINICAL TRIAL: NCT02206464
Title: VRC 315: A Phase I Open-Label, Randomized Study of H7 Influenza Prime-Boost Regimens in Healthy Adults: Recombinant H7 DNA Plasmid Vaccine, VRC-FLUDNA071-00-VP, Administered Alone or With Monovalent Influenza Subunit Virion H7N9 Vaccine (MIV) as Prime With MIV Boost Compared to MIV Prime With MIV Boost
Brief Title: H7 Influenza Prime-Boost Regimens in Healthy Adults: Recombinant H7 DNA Plasmid Vaccine, VRC-FLUDNA071-00-VP, Administered Alone or With Monovalent Influenza Subunit Virion H7N9 Vaccine (MIV) as Prime With MIV Boost Compared to MIV Prime With MIV Boo...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140160; 14-I-0160
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-01-07

CONDITIONS: Influenza
Keywords: A/Anhui/1/2013 (H7N9); Antibody Response; Avian Influenza; A/Shanghai/2/2013 (H7N9); Immunogenicity
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

ARMS (3):
- Group 1 (Experimental): H7 DNA vaccine on Day 0 and H7N9 MIV at StudyWeek 16
  Interventions: Biological: A/Shanghai/02/2013 (H7N9) MIV; Biological: VRC-FLUDNA071-00-VP
- Group 2 (Experimental): H7 DNA and H7N9 MIV administered on Day 0 and H7N9 MIV boost at Study Week 16
  Interventions: Biological: A/Shanghai/02/2013 (H7N9) MIV; Biological: VRC-FLUDNA071-00-VP
- Group 3 (Experimental): H7N9 MIV on Day 0 and H7N9 MIV at Study Week 16
  Interventions: Biological: A/Shanghai/02/2013 (H7N9) MIV; Biological: VRC-FLUDNA071-00-VP

INTERVENTIONS:
Biological: A/Shanghai/02/2013 (H7N9) MIV — Monovalent Influenza Subvirion Vaccine for H7N9 avian influenza (H7N9 MIV)
Biological: VRC-FLUDNA071-00-VP — H7 DNA Vaccine

SUMMARY:
Background:<TAB>

- Flu virus that causes disease in birds can sometimes spread to people. It can cause severe illness, even death. Vaccines are used to try to create resistance to such infections. Researchers want to test a new vaccination strategy, combining two different vaccine types, the H7 DNA Vaccine (DNA vaccine) and H7N9 Monovalent Inactivated Vaccine (MIV), to see if one of two combinations offer better protection against a certain type of bird flu in humans when compared to vaccination using two doses of MIV alone.

Objectives:

* To see if 2 vaccines for bird flu, are safe and tolerable for humans.
* To study immune responses to these vaccines.

Eligibility:

- Healthy adults 18 60 years old.

Design:

* Participants will be screened through a separate protocol.
* Participants will be randomly assigned to 1 of 3 groups. Each group will get a different combination of vaccines.
* Participants will have about 8 clinic visits. Each visit takes 2 4 hours. Blood will be drawn at some visits. Urine samples may be collected.
* Participants will receive vaccinations at 2 of the visits, 16 weeks apart.
* The H7N9 MIV will be injected in the upper arm using a needle and syringe. The DNA vaccine will be injected in the upper arm using a device that delivers the vaccine through the skin by pressure instead of a needle.
* Participants will be observed for at least 30 minutes after each vaccination.
* Soon after each vaccination, participants will get 1 2 phone calls, come to clinic for evaluation, and complete a diary at home for 1 week. They will record their temperature and symptoms and look at the injection site daily.
* Participants will have follow-up blood tests.

DETAILED DESCRIPTION:
VRC 315 STUDY:

A Phase I Open-Label, Randomized Study of H7 Influenza Prime-Boost Regimens in Healthy Adults: Recombinant H7 DNA Plasmid Vaccine, VRC-FLUDNA071-00-VP, Administered Alone or with Monovalent Influenza Subunit Virion H7N9 Vaccine (MIV) as Prime with MIV Boost Compared to MIV Prime with MIV Boost

STUDY DESIGN:

This is a Phase I, randomized, open-label study to evaluate the safety, tolerability, and immunogenicity of prime-boost vaccination regimens against H7N9 Influenza. A vaccination regimen with the VRC-FLUDNA071-00-VP (H7 DNA) vaccine administered alone or concurrently in different arms with A/Shanghai/2/2013(H7N9) (MIV) as prime followed by inactivated MIV boost will be compared to MIV-MIV prime-boost with a 16 week boost interval. The primary hypothesis is that all the H7 DNA prime-MIV boost, DNA+MIV prime-MIV boost, and MIV-MIV study regimens will be safe for human administration. A secondary hypothesis is that the H7 DNAMIV regimen will elicit a greater frequency and/or magnitude of antibody against H7 than the MIV-MIV regimen. The primary objective is to evaluate the safety and tolerability in healthy adults of the investigational vaccine regimens. Secondary objectives are related to the immunogenicity of the vaccination regimens.

PRODUCT DESCRIPTION:

The investigational VRC-FLUDNA071-00-VP vaccine was developed by VRC, NIAID and is composed of a single closed-circular DNA plasmid that encodes the H7 hemagglutinin (HA) protein of A/Anhui/1/2013 (H7N9) influenza, and is supplied in single dose vials at a concentration of 4 mg/mL. H7 DNA vaccinations will be 4 mg administered as a 1 mL intramuscularly (IM) using the Biojector o 2000 Needle-Free Injection Management System (Biojector). The inactivated H7N9 vaccine is monovalent subunit virion vaccine, A/Shanghai/2/2013(H7N9) MIV, manufactured by Sanofi Pasteur, Inc (Swiftwater, PA), and supplied at 30 mcg/0.5 mL per vial. The H7N9 MIV vaccinations will be 45 mcg administered as a 0.75 mL IM injection using needle and syringe. All injections will be in the deltoid muscle.

SUBJECTS:

A total of up to 36 healthy adults, ages 18-60 years will be enrolled.

STUDY PLAN:

Subjects will be randomized equally into the three study groups and will receive two vaccinations as shown in the schema. The protocol requires 7 clinic visits and a telephone follow-up contact after each study injection. Durability of immune response will be followed through Study Week 28.

STUDY DURATION:

Subjects will be evaluated for safety and immune responses throughout the study for 12 weeks following the boost. Duration of time on study will be 28 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

1. 18 to 60 years old.
2. Available for clinic visits for up to 28 weeks after enrollment.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Willing to donate blood for sample storage to be used for future research.
5. In good general health without clinically significant medical history.
6. Received a current seasonal influenza vaccine at least 2 weeks before enrollment.
7. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 56 days prior to enrollment.

   Laboratory Criteria within 56 days prior to enrollment:
8. Hemoglobin within institutional normal limits
9. White blood cells (WBC) and differential either within institutional normal range or accompanied by site physician approval
10. Total lymphocyte count greater than or equal to 800 cells/mm3
11. Platelets = 125,000 500,000/mm3
12. Alanine aminotransferase (ALT) less than or equal to 1.25 x upper limit of normal (ULN)
13. Serum creatinine less than or equal to .1 x ULN based on the institutional normal range

    Criteria applicable to women of childbearing potential:
14. Negative human chorionic gonadotropin ( <=-HCG) pregnancy test (urine or serum) on day of enrollment
15. Agree to use an effective means of birth control from 21 days prior to enrollment through 4 weeks after the second study vaccination

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply. Women Specific:

1. Breast-feeding or planning to become pregnant while participating in the study

   Subject has received any of the following substances:
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
3. Blood products within 16 weeks prior to enrollment
4. Live attenuated vaccines within 4 weeks prior to initial study vaccine administration
5. Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
6. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal within 2 weeks of initial study vaccine administration unless approved by the study Principal Investigator (PI)
7. Allergy treatment with antigen injections, unless on maintenance schedule
8. Current anti-TB prophylaxis or therapy
9. Previous H7 avian influenza investigational vaccine

   Subject has a history of any of the following clinically significant conditions:
10. Contraindication to receiving an FDA-approved current seasonal influenza vaccination including hypersensitivity to eggs
11. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator
12. Hereditary angioedema, acquired angioedema, or idiopathic forms of Angioedema
13. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes
15. Thyroid disease that is not well controlled
16. Idiopathic urticaria within the past year
17. Hypertension that is not well controlled
18. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study
20. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Type 1 hypersensitivity reaction to aminoglycoside antibiotics
23. Guillain-Barr(SqrRoot)(Copyright) Syndrome
24. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt
25. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07-29; Primary Completion 2016-01-07 (Actual); Study Completion 2016-01-07 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events (reactogenicity). | Daily for 7 days following each vaccination.
Adverse events of all severities. | Through 28 days after each injection.
Serious adverse events, new chronic medical conditions and influenza-like illnesses | From first vaccination to last study visit

SECONDARY OUTCOMES:
H7-specific antibody response as measured by HAI assay | Day 0 (baseline) and 2 weeks after the boost vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ledgerwood JE, Graham BS. DNA vaccines: a safe and efficient platform technology for responding to emerging infectious diseases. Hum Vaccin. 2009 Sep;5(9):623-6. doi: 10.4161/hv.8627. No abstract available. PMID 19779298
- [Background] Ledgerwood JE, Wei CJ, Hu Z, Gordon IJ, Enama ME, Hendel CS, McTamney PM, Pearce MB, Yassine HM, Boyington JC, Bailer R, Tumpey TM, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 306 Study Team. DNA priming and influenza vaccine immunogenicity: two phase 1 open label randomised clinical trials. Lancet Infect Dis. 2011 Dec;11(12):916-24. doi: 10.1016/S1473-3099(11)70240-7. Epub 2011 Oct 3. PMID 21975270
- [Background] Ledgerwood JE, Zephir K, Hu Z, Wei CJ, Chang L, Enama ME, Hendel CS, Sitar S, Bailer RT, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 310 Study Team. Prime-boost interval matters: a randomized phase 1 study to identify the minimum interval necessary to observe the H5 DNA influenza vaccine priming effect. J Infect Dis. 2013 Aug 1;208(3):418-22. doi: 10.1093/infdis/jit180. Epub 2013 Apr 30. PMID 23633407